CLINICAL TRIAL: NCT05338255
Title: Evaluation of the Clinical Pathway of Intensified Recovery Surgery for Adults in the Processes of Total Knee and Hip Replacement at the Maz Hospital
Brief Title: Results of the Application of the Clinical Pathway of Intensified Recovery Surgery for Adults in the Processes of Total Knee and Hip Replacement at the Maz Hospital
Status: Completed | Type: Observational
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Silvia Gomez Gomez, Principal Investigator, Universidad de Zaragoza
Other Study IDs: Silvia Gómez Gómez
Record Dates: First submitted 2022-04-13; First posted 2022-04-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Arthropathy of Knee; Arthropathy of Hip
Keywords: Arthroplasty; Fast-track surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who have undergone surgery at the MAZ hospital for knee/hip replacement.

SUMMARY:
The investigators are going to study all the patients who have undergone surgery at the MAZ hospital from 2019 to the present for knee replacement and hip replacement. The investigators want to analyze the results to see if applying the RICA clinical pathway results are better.

ELIGIBILITY:
Inclusion Criteria:

* Adults, over 18 years old.
* Diagnosis of moderate-severe gonarthrosis or moderate-severe coxarthrosis.
* Patients who are operated by orthopedic surgeons at MAZ Hospital with knee or hip arthroplasty.
* Between January 2019 and June 2022.
* ASA I-II-III.

Exclusion Criteria:

* ASA IV.
* Minors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People who is attended at MAZ Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 534 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Degree of compliance with the criteria for performing surgery according to the clinical pathway | One month postoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Silvia Gómez Gómez, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No